CLINICAL TRIAL: NCT04299672
Title: Effect of Postural Reconstruction on the Functionality of the Cervical Region
Brief Title: Cervical Functionality and Posture (CERFUPOS)
Acronym: CERFUPOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Antonio de Nebrija (Other)
Responsible Party: Principal Investigator, José Ríos-Díaz, Faculty-Reseacher, Universidad Antonio de Nebrija
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR_Cervical
Record Dates: First submitted 2019-11-01; First posted 2020-03-09 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: People With Impaired Motor Function in the Cervical Region
Keywords: Cervical pain; Funcionality; Posture; Balance; Muscular tone; Postural reconstruction; Physical Therapy
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: One group
Masking Description: Therapist and outcome assessors are independent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postural reconstruction (Experimental): Maximum external rotation of the hip in lower limb elevation and the dorsal flexion of the ankle with flexion of the toes, performed in both lower limbs alternately and independent.
  Participant must control breathing. The detail phases of a general intervention are:
  1. PASSIVE displacement of the segment until reaching CRITICAL AMPLITUDE, which corresponds to the light myofascial stress or to the appearance of evoked responses.
  2. ACTIVE MAINTENANCE of the critical amplitude.
  3. WORK BREATHING.
  4. INDUCTIVE ACTIVE APPLICATIONS with movements of great relative amplitude.
  5. FINISHING CRITERIA: reduction or extinction of evoked responses, patient fatigue or execution of the technique for 15 minutes without any of the above premises having been reached.
  Interventions: Procedure: Postural reconstruction

INTERVENTIONS:
Procedure: Postural reconstruction — Interventions are described in group descriptions

SUMMARY:
BACKGROUND: Musculoskeletal alterations of the cervical region constitute clinical situations with a high prevalence that may be related to posture mismatches. Static alterations not linked to a defined pathological picture may come from a sensory-motor disorder whose main manifestations are increased muscle tone and stiffness. Postural reconstruction (RP). The RP method has as main objective the rebalancing of the muscular tone from 1) the sensorimotor recovery and 2) the re-functionalization of the subcortical toninergic centers. The aim of this study is to determine the effect of this physiotherapeutic approach on the functionality and posture of the cervical region.

OBJECTIVES: 1) to know the effect of PR on cervical function in subjects with impaired cervical motor function; and 2) to know the effect of PR on static in subjects with impaired cervical motor function.

PARTICIPANTS & METHODS: quasi-experimental design, with only one intervention group (N=40). Data records before and after the 1st intervention, before the 2nd, 4th and 6th weekly treatment sessions, at 15 days and a month and at 3 months after the end of treatment.

INTERVENTION: The intervention will consist of the application of a RP maneuver applied to both lower limbs to obtain improvements in the cranio-cervical region.

OUTCOMES: The outcome variables will collect information on active joint movement in the cervical region, anatomical references representative of body statics, cervical repositioning, cervical disability, pain and time to extinction of the effect.

DETAILED DESCRIPTION:
SAMPLE: People between 18-45 years old and with 1) alteration of active cervical mobility in at least one of the six directions of analytic movement compared to normality or with alteration of motor control of the cervical region in at least one of the 7 tests included in the study compared to normal criteria.

SAMPLE SIZE: The minimum size required has been calculated using the program G*Power 3.1.3 for Windows (University Kiel, Germany, 2008) based on an effect size of 0.5, type I error of 5%,type II error of 10%, an effect size of delta=0.20, a intra-measures correlation =0.5 for 7 measurement points. An extra 20% for drop-outs was added. The final sample size is N=40.

INTERVENTION:

Maximum external rotation of the hip in lower limb elevation and the dorsal flexion of the ankle with flexion of the toes, performed in both lower limbs alternately and independently. During the performance of the technique, the patient must implement the work breathing learned in the first basal assessment session.

It will be applied weekly during 6 consecutive weeks.

DATA ANALYSIS:

1. -Database cleaning and out-of-range data detection using Excel validation techniques.
2. -For statistical analysis, a descriptive analysis using means and standard deviations will be performed, as well as ranges and quartiles for quantitative measurements. Qualitative variables shall be summarised by counts and frequencies. The assumption of normality (Kolmogorv-Smirnoff test) and sphericity (Maulchy's test) prior to the analysis of variance (ANOVA) will be checked for repeated measurements in which only the intra-unit factors (7 time measurements). Pair comparisons were made with the Dunn-Bonferroni correction for type I erro and the age, sex and BMI variables were entered into the model as covariates to estimate their possible effect on the dependent variables.

The percentages of change from the baseline values in the intragroup comparison shall be calculated. The effect size will be estimated with the Hedges' g statistic.

The significance level will be set to p<0.05 and calculations will be performed with jmv r package for R (R Core Team, 2019. R: A language and environment for statistical. computing. R Foundation for Statistical Computing, Vienna, Austria. URL http://www.R-project.org/)

ELIGIBILITY:
Inclusion Criteria:

* Alteration of active cervical mobility in at least one of the six directions of analytic movement compared to normality.
* Alteration of motor control of the cervical region in at least one of the 7 tests included in the study, compared with the criteria of normality.

Exclusion Criteria:

* Traumatic cervical history (whiplash, head trauma, etc.)
* Diagnosis of degenerative diseases of any origin or known cervical degenerative signs.
* Diagnosis of diseases of neurological origin or cerebrovascular alteration.
* Diagnosis of cardiovascular or respiratory disease affecting the pattern of ventilation.
* Pharmacological treatment (muscle relaxants, analgesics or anti-inflammatories) up to 4 weeks before the start of the study or during the study on a regular basis.
* Pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Change in Craniovertebral angle | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  The craniovertebral angle is defined as the angle between the line from the external auditory meatus to the seventh cervical vertebra and a horizontal line at the level of the seventh cervical vertebra. The measure will be carried out with the KINOVEA system in degrees.
Change in Sternum-mentonian distance | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  The Sternum-mentonian distance is the distance between the distal end of the mentonand the proximal end of the sternal notch. The measure will be carried out with the KINOVEA system in centimeters.
Change in Head-neck asymmetry in the frontal plane | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Head-neck asymmetry in the frontal plane is the deviation of the fronto-naso-mentonian line from the vertical line of the body axis. The measure will be carried out with the KINOVEA system in centimeters.
Change in Displacement of the center of masses | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Displacement of the center of masses by means of a Dinascan/IBV dynamometer platform with NedSVE/IB balance evaluation system.
Change in Upper cervical active rotation test | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Upper cervical active rotation on 4 supports. The correct movement pattern implies that the patient is able to dissociate the upper rotation movement.
Change in Upper cervical active flexion test | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Upper cervical active flexion on 4 supports. The correct movement pattern implies that the sagittal movement axis is correct and balanced. The normal bending movement must be "clean" and regular in the upper and lower cervical area, almost touching the sternum
Change in Active cervical extension in seating test | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Active cervical extension in seating. The correct pattern should be smooth and uniform top, middle, bottom. NO HINGES. The face line stays about 15 - 20º from the horizontal.
Change in Recover neutral position from cervical extension test | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Return to the neutral position from the active cervical extension position when seated. The correct pattern is soft starting with the cranio-cervical area and continuing with the rest of the cervical spine.
Change in Active bilateral flexion of shoulders test | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Active bilateral bending of both upper limbs in standing position. The cervical spine should remain static during the 180º of bilateral upper limb elevation.
Change in Active unilateral flexion of shoulders test | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Active unilateral bending of both upper limbs in standing position. The cervical spine should remain static during the 180º of unilateral upper limb elevation.
Change in Rear balancing on 4 supports test | Pre-intervention, immediately post-intervention, 2nd, 4th, 6th intervention, 15, 30 days post-intervention and 3 months post-intervention
  During the sitting gesture on the heels the cervical spine should be static.
Change in Cervical discapacity | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Neck disability Index. The NDI is a modification of the Oswestry Low Back Pain Disability Index . It is a patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation with a range from 0 (no activity limitations) to 50 (complete activity limitation)
Change in Cervical pain | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Numeric Pain Rating Scale in a range from 0 (no pain) to 100 (maximum pain).

SECONDARY OUTCOMES:
Change in Cervical Flexion | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Cervical flexion with goniometry (in degrees)
Change in Cervical Extension | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Cervical extension with goniometry (in degrees)
Change in Cervical Inclination | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Cervical inclination bilaterally with goniometry (in degrees).
Change in Cervical Rotation | Pre-intervention, immediately after first intervention, post-2nd-intervention(2 weeks), post-4th-intervention (4 weeks), post-6th-intervention (6 weeks) and follow-up at 15 days, 30 days and 3 months
  Cervical rotation bilaterally with goniometry (in degrees).

CONTACTS AND LOCATIONS:
Locations (1):
- José Ríos-Díaz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fejer R, Kyvik KO, Hartvigsen J. The prevalence of neck pain in the world population: a systematic critical review of the literature. Eur Spine J. 2006 Jun;15(6):834-48. doi: 10.1007/s00586-004-0864-4. Epub 2005 Jul 6. PMID 15999284
- [Background] Sempere-Rubio N, Aguilar-Rodriguez M, Espi-Lopez GV, Cortes-Amador S, Pascual E, Serra-Ano P. Impaired Trunk Posture in Women With Fibromyalgia. Spine (Phila Pa 1976). 2018 Nov 15;43(22):1536-1542. doi: 10.1097/BRS.0000000000002681. PMID 29652782
- [Background] Kim EK, Kim JS. Correlation between rounded shoulder posture, neck disability indices, and degree of forward head posture. J Phys Ther Sci. 2016 Oct;28(10):2929-2932. doi: 10.1589/jpts.28.2929. Epub 2016 Oct 28. PMID 27821964
- [Background] Kim JY, Kwag KI. Clinical effects of deep cervical flexor muscle activation in patients with chronic neck pain. J Phys Ther Sci. 2016 Jan;28(1):269-73. doi: 10.1589/jpts.28.269. Epub 2016 Jan 30. PMID 26957772
- [Background] Griegel-Morris P, Larson K, Mueller-Klaus K, Oatis CA. Incidence of common postural abnormalities in the cervical, shoulder, and thoracic regions and their association with pain in two age groups of healthy subjects. Phys Ther. 1992 Jun;72(6):425-31. doi: 10.1093/ptj/72.6.425. PMID 1589462
- [Background] Ferracini GN, Chaves TC, Dach F, Bevilaqua-Grossi D, Fernandez-de-Las-Penas C, Speciali JG. Relationship Between Active Trigger Points and Head/Neck Posture in Patients with Migraine. Am J Phys Med Rehabil. 2016 Nov;95(11):831-839. doi: 10.1097/PHM.0000000000000510. PMID 27149581
- [Background] Malmstrom EM, Olsson J, Baldetorp J, Fransson PA. A slouched body posture decreases arm mobility and changes muscle recruitment in the neck and shoulder region. Eur J Appl Physiol. 2015 Dec;115(12):2491-503. doi: 10.1007/s00421-015-3257-y. Epub 2015 Oct 1. PMID 26429723
- [Background] Janda V. On the concept of postural muscles and posture in man. Aust J Physiother. 1983 Jun;29(3):83-4. doi: 10.1016/S0004-9514(14)60665-6. PMID 25025491
- [Background] Wilke J, Krause F, Vogt L, Banzer W. What Is Evidence-Based About Myofascial Chains: A Systematic Review. Arch Phys Med Rehabil. 2016 Mar;97(3):454-61. doi: 10.1016/j.apmr.2015.07.023. Epub 2015 Aug 14. PMID 26281953
- [Background] Krause F, Wilke J, Vogt L, Banzer W. Intermuscular force transmission along myofascial chains: a systematic review. J Anat. 2016 Jun;228(6):910-8. doi: 10.1111/joa.12464. Epub 2016 Mar 22. PMID 27001027
- [Background] Destieux C, Gaudreault N, Isner-Horobeti ME, Vautravers P. Use of Postural Reconstruction(R) physiotherapy to treat an adolescent with asymmetric bilateral genu varum and idiopathic scoliosis. Ann Phys Rehabil Med. 2013 May;56(4):312-26. doi: 10.1016/j.rehab.2013.02.004. Epub 2013 Mar 20. PMID 23541175
- [Background] Weiler C, Schietzsch M, Kirchner T, Nerlich AG, Boos N, Wuertz K. Age-related changes in human cervical, thoracal and lumbar intervertebral disc exhibit a strong intra-individual correlation. Eur Spine J. 2012 Aug;21 Suppl 6(Suppl 6):S810-8. doi: 10.1007/s00586-011-1922-3. Epub 2011 Aug 12. PMID 21837413
- [Background] Christe A, Laubli R, Guzman R, Berlemann U, Moore RJ, Schroth G, Vock P, Lovblad KO. Degeneration of the cervical disc: histology compared with radiography and magnetic resonance imaging. Neuroradiology. 2005 Oct;47(10):721-9. doi: 10.1007/s00234-005-1412-6. Epub 2005 Sep 1. PMID 16136264
- [Result] Czaprowski D, Stolinski L, Tyrakowski M, Kozinoga M, Kotwicki T. Non-structural misalignments of body posture in the sagittal plane. Scoliosis Spinal Disord. 2018 Mar 5;13:6. doi: 10.1186/s13013-018-0151-5. eCollection 2018. PMID 29516039
- [Result] Pausic J, Pedisic Z, Dizdar D. Reliability of a photographic method for assessing standing posture of elementary school students. J Manipulative Physiol Ther. 2010 Jul-Aug;33(6):425-31. doi: 10.1016/j.jmpt.2010.06.002. PMID 20732579
- [Result] Rosario JL. Biomechanical assessment of human posture: a literature review. J Bodyw Mov Ther. 2014 Jul;18(3):368-73. doi: 10.1016/j.jbmt.2013.11.018. Epub 2013 Nov 27. PMID 25042306
- [Result] Fortin C, Feldman DE, Cheriet F, Labelle H. Clinical methods for quantifying body segment posture: a literature review. Disabil Rehabil. 2011;33(5):367-83. doi: 10.3109/09638288.2010.492066. Epub 2010 Jun 23. PMID 20568973
- [Result] Guan X, Fan G, Wu X, Zeng Y, Su H, Gu G, Zhou Q, Gu X, Zhang H, He S. Photographic measurement of head and cervical posture when viewing mobile phone: a pilot study. Eur Spine J. 2015 Dec;24(12):2892-8. doi: 10.1007/s00586-015-4143-3. Epub 2015 Jul 24. PMID 26206292
- [Result] Cernean N, Serranheira F, Goncalves P, Sa Dos Reis C. Ergonomic strategies to improve radiographers' posture during mammography activities. Insights Imaging. 2017 Aug;8(4):429-438. doi: 10.1007/s13244-017-0560-7. Epub 2017 Jun 21. PMID 28639113
- [Result] Segarra V, Duenas L, Torres R, Falla D, Jull G, Lluch E. Inter-and intra-tester reliability of a battery of cervical movement control dysfunction tests. Man Ther. 2015 Aug;20(4):570-9. doi: 10.1016/j.math.2015.01.007. Epub 2015 Jan 26. PMID 25677675
- [Result] Luomajoki H, Kool J, de Bruin ED, Airaksinen O. Movement control tests of the low back; evaluation of the difference between patients with low back pain and healthy controls. BMC Musculoskelet Disord. 2008 Dec 24;9:170. doi: 10.1186/1471-2474-9-170. PMID 19108735
- [Result] Revel M, Andre-Deshays C, Minguet M. Cervicocephalic kinesthetic sensibility in patients with cervical pain. Arch Phys Med Rehabil. 1991 Apr;72(5):288-91. PMID 2009044
- [Result] Roren A, Mayoux-Benhamou MA, Fayad F, Poiraudeau S, Lantz D, Revel M. Comparison of visual and ultrasound based techniques to measure head repositioning in healthy and neck-pain subjects. Man Ther. 2009 Jun;14(3):270-7. doi: 10.1016/j.math.2008.03.002. Epub 2008 Jun 2. PMID 18514016
- [Result] Kovacs FM, Bago J, Royuela A, Seco J, Gimenez S, Muriel A, Abraira V, Martin JL, Pena JL, Gestoso M, Mufraggi N, Nunez M, Corcoll J, Gomez-Ochoa I, Ramirez MJ, Calvo E, Castillo MD, Marti D, Fuster S, Fernandez C, Gimeno N, Carballo A, Milan A, Vazquez D, Canellas M, Blanco R, Brieva P, Rueda MT, Alvarez L, Del Real MT, Ayerbe J, Gonzalez L, Ginel L, Ortega M, Bernal M, Bolado G, Vidal A, Ausin A, Ramon D, Mir MA, Tomas M, Zamora J, Cano A. Psychometric characteristics of the Spanish version of instruments to measure neck pain disability. BMC Musculoskelet Disord. 2008 Apr 9;9:42. doi: 10.1186/1471-2474-9-42. PMID 18400084
- [Result] Young IA, Dunning J, Butts R, Cleland JA, Fernandez-de-Las-Penas C. Psychometric properties of the Numeric Pain Rating Scale and Neck Disability Index in patients with cervicogenic headache. Cephalalgia. 2019 Jan;39(1):44-51. doi: 10.1177/0333102418772584. Epub 2018 Apr 19. PMID 29673262